CLINICAL TRIAL: NCT05915390
Title: Effects of Walnuts on Innate, Acquired and Gut Immunity in Older Adults With Overweight: A Randomized Controlled Trial
Brief Title: Walnut and Immunity Study
Acronym: walnutimmune
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor Nutrition and Epidemiology, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5220423
Record Dates: First submitted 2023-05-16; First posted 2023-06-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Immune Response; Upper Respiratory Tract Infection
Keywords: walnuts; Immunity; Inflammation
MeSH Terms: conditions — Respiratory Tract Infections; Inflammation

STUDY DESIGN:
Intervention Model Description: This will be a parallel, free-living, randomized controlled trial with 54 men and post-menopausal women
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will not be aware which participant is in what arm. The participant and the care provider will know about the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walnut group (Active Comparator): walnut group will receive 15% of their total energy as walnuts
  Interventions: Dietary Supplement: walnuts
- control group (Active Comparator): continue with habitual diet and abstain from eating walnuts
  Interventions: Dietary Supplement: Habitual diet

INTERVENTIONS:
Dietary Supplement: walnuts — walnuts will provide 15% of the total energy
  Arms: walnut group
Dietary Supplement: Habitual diet — continue with habitual diet and abstain from walnuts
  Arms: control group

SUMMARY:
The main objective of the study is to determine if eating walnuts enhances immune function, in older free-living men and postmenopausal women with overweight.

DETAILED DESCRIPTION:
The main objectives of our proposed study are to determine the effect of walnut consumption on innate, acquired, and gut immunity by assessing whether the ingestion of walnuts enhances immune function, in older free-living men and postmenopausal women with overweight. To accomplish these objectives, a randomized controlled, parallel design study is proposed with two groups consuming their habitual diet, but with one (Walnut group) receiving 15% of their total energy as walnuts and the other (Control group) abstaining from eating any walnuts and limited amounts of other tree nuts and peanuts (up to <1 serving/wk).

ELIGIBILITY:
Inclusion Criteria:

* Older men and post-menopausal women aged 55-75 years
* Have a BMI of 25-32
* Being able to commute to Loma Linda University.
* Not taking medication or supplements that affect immunity

Exclusion Criteria:

* Intolerance or allergy to walnuts
* Regular intake of walnuts and/or other nuts (>3 ounces per week).
* Immune system insufficiency or disease.
* Using immune boosting supplements.
* Exposure to antibiotics and corticoids immediately prior to the study.
* Participants with uncontrolled chronic diseases, and relevant psychiatric illness, including major depression will not be included in study
* Flu vaccination or Covid booster within past 6 months

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
changes in lymphocyte populations | baseline to 12 weeks
  Immunophenotyping will be performed by flow cytometry to measure the number of T helper, T cytotoxic, Naïve and memory cells and B cells
changes in lymphocyte activity | baseline to 12 weeks
  The production of lymphocytes will be measured in the supernatant using Enzyme linked immunosorbent assay (ELISA)
changes in cytokine production | baseline to 12 weeks
  The cytokines produced due to lymphocyte activity will be measured in the supernatant using Enzyme linked immunosorbent assay (ELISA)
changes in serum inflammatory cytokine concentration | baseline to 12 weeks
  changes in the concentrations of the inflammatory cytokines will be performed on serum using enzyme-linked immunoassay (ELISA) will include hs-CRP, interleukin (IL)-1β, IL-6, TNF-α, IL-10, and IL-4.
changes in diversity of immune-modulating and butyrate -producing gut bacteria in feces | baseline to 12 weeks
  DNA extraction from stool samples will be performed using QIAamp DNA Stool Mini kits.69 The QIIME (Quantitative Insights Into Microbial Ecology) software will be used to analyze 16S rRNA gene sequences and determine the effect of the intervention on microbial diversity at the phylum, genus, and operational taxonomic unit levels.
Changes in concentration of Immunoglobulin A in feces | baseline to 12 weeks
  changes in Immunoglobulin A will be determined using high performance liquid chromatography-mass spectrometry (HPLC-MS)
Changes in concentration of Calprotectin in feces | baseline to 12 weeks
  changes in Calprotectin will be determined using high performance liquid chromatography-mass spectrometry (HPLC-MS)
Changes in concentration of small chain fatty in feces | baseline to 12 weeks
  changes in Small chain fatty acids will be determined using high performance liquid chromatography-mass spectrometry (HPLC-MS)

SECONDARY OUTCOMES:
changes in upper respiratory infection questionnaire score | baseline to 12 weeks
  Upper respiratory tract infections will be tracked using the Jackson and Dowling questionnaire. The questionnaire will be completed daily by participants, either manually or electronically , throughout the 12-week study period. The scale for the questionnaire is from 0-42. The higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No